CLINICAL TRIAL: NCT02610244
Title: Examining Benefits of Modified Cogmed Training With ADHD Youth at Cambridge Memorial Hospital (CMH)
Brief Title: Examining Benefits of Modified Cogmed Training With ADHD at Cambridge Memorial Hospital(CMH)
Acronym: CMH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original sponsor withdrew funding.
Sponsor: Cambridge Memorial Hospital (Other)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADHD-MCT-09092015; 2015-0563 (Other: Tri-Hospital Research Ethics Board); 20679 (Other: University of Waterloo Ethics)
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment As Usual (No Intervention): Standard treatment as usual as directed by the physician.
- Modified Cogmed Training (Experimental): 10 weeks of computerized training (3x weekly for 35-minutes each session) that targets thinking skills that are often impaired in individuals diagnosed with ADHD.
  Interventions: Other: Modified Cogmed Training

INTERVENTIONS:
Other: Modified Cogmed Training — Comparison of outcome measures between treatment-as-usual group and Modified Cogmed Training group after 10 weeks and 3 months follow up.
  Arms: Modified Cogmed Training

SUMMARY:
ADHD youth (8-16 years) will be randomized to either treatment-as-usual group or a modified version of the Cogmed program (MCT) that is suitable for use in a hospital setting (duration = 3 daily 35-min sessions for 10 weeks). The main objectives are to determine whether there is improvement in working memory and attention, a reduction in concerns related to ADHD and social emotional behaviour,and transfer effects for reading and math following participation in our MCT.

DETAILED DESCRIPTION:
The Cogmed working memory training program consists of 5 daily 50-min sessions for 5 weeks. This program has been identified as a promising intervention for youth with Attention Deficit Hyperactivity Disorder (ADHD) who have deficits in aspects of executive functioning (EF), such as working memory (WM) and attention (ATT), as well as social-emotional behavior (SEB). Findings regarding the efficacy and generalization of transfer effects associated with Cogmed have been mixed, possibly due to methodological limitations of the standard program. In our study, these limitations will be addressed with ADHD youth (8-16 years) in a randomized controlled trial using a modified version of the Cogmed program (MCT) that is suitable for use in a hospital setting (duration = 3 daily 35-min sessions for 10 weeks). The main objective is to determine whether there is improvement in WM and ATT, a reduction in concerns related to ADHD and SEB, and transfer effects for reading and math following participation in our MCT.

ELIGIBILITY:
Inclusion Criteria:

1. Youth who are between 8-16 years age.
2. Youth with a primary diagnosis of ADHD per psychiatric and psychological assessment.
3. Youth with an estimated Intelligence Quotient (IQ) equal or greater than 80 on an intelligence measure (Wechsler Abbreviated Scale of Intelligence; WASI), where the average IQ varies from 90-110.
4. Youth with reading comprehension at or above a grade 2 level on a standardized reading test (Wechsler Individual Achievement Test - 3rd Edition; WIAT-III).
5. Youth who are receiving medication will have made an adequate adjustment to their medication as shown by stable blood levels, psychiatric consultation, and self and parent report at least 2 weeks prior to the start of their acceptance into this study.

Exclusion Criteria:

1. Youth who are younger than 8 or older than 16 at the time of enrollment.
2. Youth who do not have a primary diagnosis of ADHD.
3. Youth with an estimated Intelligence Quotient (IQ) below 80 on an intelligence measure (Wechsler Abbreviated Scale of Intelligence; WASI), where the average IQ varies from 90-110. Children with intellectual functioning below this level have been found to have trouble following instructions that are necessary for the training program.
4. Youth with reading comprehension below a grade 2 level on a standardized reading test (Wechsler Individual Achievement Test - 3rd Edition; WIAT-III). Children with reading skills below this level have been found to have trouble following instructions that are necessary for the training program.
5. Youth do not intend to begin new medication, discontinue existing medication, or change dose in medication - unless indicated per their doctor's instructions - for the duration of their involvement in the study.
6. Youth cannot be accepted into the study if they have a significant medical impairment that would preclude their participation, a significant uncorrected visual/hearing deficit that would make it difficult for them to see a computer screen and follow verbal instructions, and/or a significant problem with their fine motor control that would make it difficult for them to use a keyboard.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes assessed for Working Memory Index (BRIEF measure) and working memory (verbal and Visual-spatial) as measured on Alloway Working Memory Test | Baseline,10 weeks, 3 months
  The BRIEF Parent/Teacher ratings of youth's working memory index and Youth 's scores on Alloway Working Memory test at baseline will be compared with scores after 10 weeks modified cogmed training or treament-as-usual, and after 3 months
Changes assessed on Beck Self-Concept | Baseline,10 weeks, 3 months
  Self-concept measures will be compared from baseline to after completing Cogmed training and at 3 month follow up.
Change assessed on Tova Attention Performance Index | Baseline,10 weeks, 3 months
  Attention Performance Index measures will be compared from baseline to after completing Cogmed training and at 3 month follow up.
Change assessed on Wiat-111 Reading comprehension and math problem-solving | Baseline,10 weeks, 3 months
  Reading Comprehension and Math problem-solving measures will be compared from baseline to after completing Cogmed training and at 3 month follow up.
Change assessed on Achenbach Reduction in Total Problems Scale | Baseline,10 weeks, 3 months
  Total Problem scale measures will be compared from baseline to after completing Cogmed training and at 3 month follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Mental Health,, Cambridge, Ontario, Canada